CLINICAL TRIAL: NCT07288554
Title: A Randomized, Double-Blind, Placebo-controlled, Single- and Multiple-ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, Pharmacodynamics and Clinical Activity of BBT002 in Healthy Volunteers and Participants With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study of BBT002 in Healthy Volunteers (HVs) and in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bambusa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BBT002-002
Record Dates: First submitted 2025-12-16; First posted 2025-12-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A Single Ascending Dose BBT002 (Experimental): A single dose of BBT002 will be administered in healthy volunteers
  Interventions: Drug: BBT002
- Part B Multiple Ascending Dose BBT002 (Experimental): Two doses of BBT002 will be administered in patients with COPD.
  Interventions: Drug: BBT002
- Part A Single Ascending Dose Placebo (Placebo Comparator): A single dose of Placebo will be administered in healthy volunteers.
  Interventions: Drug: Placebo
- Part B Multiple Ascending Dose Placebo (Placebo Comparator): Two doses of Placebo will be administered in patients with COPD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BBT002 — BBT002 will be administered
  Arms: Part A Single Ascending Dose BBT002; Part B Multiple Ascending Dose BBT002
Drug: Placebo — Placebo will be administered
  Arms: Part A Single Ascending Dose Placebo; Part B Multiple Ascending Dose Placebo

SUMMARY:
This study is a randomized, double-Blind, placebo-controlled, Single- and Multiple-ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, Pharmacodynamics and Clinical Activity of BBT002 in Healthy Volunteers and Participants with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
The study consists of two parts:

* Part A (single dose in HVs in sequential ascending dose cohorts, SAD in HVs part)
* Part B (two repeated doses in patients with COPD, MAD in patients part)

ELIGIBILITY:
Inclusion Criteria:( A&B)

1. Age of 18-65 years (HVs), 35-75 years (patients)
2. Body mass index between 18-32 kg/m², capped at 120 kg
3. Negative pregnancy tests for women of childbearing potential
4. Willingness to refrain from alcohol consumption for 24 hours prior to each study visit
5. Non-smokers, healthy current smokers (≤5 cigarettes/day), or ex-smokers
6. Adequate contraception use (for men and women of childbearing potential)
7. No clinically significant abnormalities or history of relevant diseases

Key Inclusion Criteria (Part B only)

1. Documented history of COPD with a post-bronchodilator FEV1/FVC < 0.70
2. FEV1 ≥ 50% and FEV1<80% predicted at screening.

Exclusion Criteria:( part A & B)

1. Positive viral serology for human immunodeficiency virus (HlV), hepatitis C virus (HCV), or hepatitis B (HBV)
2. Immunodeficiencies, autoimmune diseases, or cancer, history of conditions predisposing to infections
3. History of major metabolic, dermatological, liver, kidney, hematological or other significant disorders
4. Clinically relevant abnormal lab results, including low blood counts, liver enzymes, or abnormal kidney function
5. Positive drug/alcohol tests or abnormal vital signs at screening or Day -1
6. Abnormal Electrocardiogram(ECG) findings
7. History of drug/alcohol abuse in the past 2 years
8. History of severe allergic reactions or hypersensitivity

Key Exclusion Criteria for (Part B only)

1. Current diagnosis of other significant pulmonary disease
2. Significant or unstable cardiovascular diseases
3. Recent clinically significant infection
4. Inability to perform spirometry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events following single and multiple administration of BBT002 | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  Incidence, relatedness, and severity of adverse events (AEs) graded per CTCAE v5.0.
Number of participants with change in Laboratory assessments | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  Laboratory assessments include hematology, coagulation, clinical chemistry and urinalysis
Number of participants with change in vital sign measurements following dose administration. | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  Blood pressure and heart rate will be assessed.
Number of participants with change in physical examination following dose administration. | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  Physical examination will be assessed.
Number of participants with change in 12-lead ECG readings | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  12-lead ECG will be assessed.

SECONDARY OUTCOMES:
PK parameters- maximum observed concentration (Cmax) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Maximum observed concentration of the study drug in serum will be analyzed for all subjects
PK parameters- Time for maximum observed Concentration (Tmax) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Serum PK Tmax will be analyzed for all subjects
PK parameters- Area under the curve (AUC) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Area under the curve of the study drug in serum will be analyzed for all subjects
PK parameters- Volume of distribution (Vz) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Volume of distribution of the study drug in serum will be analyzed for all subjects
PK parameters- Total clearance (CL) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Total clearance of the study drug in serum will be analyzed for all subjects
PK parameters- - Elimination Half-life (t1/2) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Elimination half-life of the study drug in serum will be analyzed for all subjects
The immunogenicity of BBT002 is measured as the number and percentage of subjects who develop Anti-Drug Antibodies (ADA). | At specified timepoints pre-dose and up to 169 days post first dose administration
  Serum Anti-Drug Antibodies will be analyzed for all subject

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - The Second Hospital of Anhui Medical Univesity, Hefei, Anhui
  - The third affiliated hosptial of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Medical University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - The First People's Hospital of Xinxiang City, Xinxiang, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Chengdu fifth People's Hospital, Chengdu, Sichuang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang